CLINICAL TRIAL: NCT04084353
Title: Evaluating the Impact of Introducing a Two Stage Intrapartum Fetal Monitoring Assessment Using Intermittent Auscultation and Cardiotocography in a Government Hospital, Nagpur, India
Brief Title: Evaluating a Two Stage Intrapartum Fetal Assessment in India
Status: Completed | Type: Observational
Sponsor: University of Liverpool (Other)
Collaborators: Government Medical College, Nagpur (Industry); Gynuity Health Projects (Other)
Responsible Party: Principal Investigator, Andrew D Weeks, Professor of International Maternal Health, University of Liverpool
Other Study IDs: 4835
Record Dates: First submitted 2019-07-26; First posted 2019-09-10 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Intrapartum Fetal Monitoring
Keywords: intra partum fetal monitoring; training; quality improvement; intermittent cardiotocography (CTG); intermittent auscultation; perinatal outcomes; caesarean section rate; obstetric outcomes; India

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Delivered women: Maternal and perinatal outcomes will be collected prospectively on all patients that deliver in Government Medical College (GMC) Hospital before, during and after the training over the study period (8 months) in order to evaluate the impact of the training.
  Interventions: Other: Intrapartum fetal monitoring training and quality improvement project

INTERVENTIONS:
Other: Intrapartum fetal monitoring training and quality improvement project — Intrapartum fetal monitoring training

SUMMARY:
An intrapartum fetal monitoring training programme (on intermittent auscultation and cardiotocography) will be delivered at Government Medical College (GMC) to all relevant staff. This quality improvement project and training evaluation aims to assess and evaluate the impact of this training. This will allow the investigators to understand if it is feasible and acceptable to staff, increases knowledge and improves patient outcomes.

DETAILED DESCRIPTION:
As part of Misoprostol or Oxytocin for Labour Induction (MOLI) randomised controlled trial (RCT) (CTRI no. NCT03749902), Government Medical College (GMC) plans to increase the number of cardiotocography (CTG) machines available on labour ward and provide a United Kingdom (UK) based obstetrician to deliver training on cardiotocography (CTG) interpretation in order to improve fetal monitoring for this high risk population.

An intrapartum fetal monitoring training programme (on intermittent auscultation and cardiotocography) will be delivered at Government Medical College (GMC) to all relevant staff. This quality improvement project and training evaluation aims to assess and evaluate the impact of this training. This will allow the investigators to understand if it is feasible and acceptable to staff, increases knowledge and improves patient outcomes. It will be done through staff questionnaires, pre-and-post test scores and by examining the effects on maternal and perinatal outcomes using Kirkpatrick's training evaluation.

The whole project aims:

* To understand current practice and maternal and perinatal outcomes in Government Medical College (GMC)
* To improve intrapartum fetal monitoring with intermittent auscultation and cardiotocography (CTG)
* To improve perinatal morbidity and mortality rates
* To reduce caesarean section rates for presumed fetal compromise

ELIGIBILITY:
Inclusion Criteria:

* All women that deliver within the obstetrics department in Government Medical College (GMC) during the study period (8 months)

Exclusion criteria:

* Deliveries in A&E/medical wards
* Home deliveries
* Patients delivered in other hospitals/ambulance deliveries
* Macerated still birth
* Fresh still birth with no fetal heart on admission to hospital

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women delivered in Government Medical College (GMC) Hospital, Nagpur, India, over two months before, during and two months after project implementation
Study Population: All women that deliver within the obstetrics department in Government Medical College (GMC) during the study period (8 months)
Sampling Method: Non-Probability Sample
Enrollment: 6682 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Caesarean section performed for presumed fetal compromise as a prortion of all caesarean sections | 8 months
  Percentage change of rate per month

SECONDARY OUTCOMES:
Intrapartum fetal monitoring - Improved documentation | 8 months
  Average number of times fetal heart rate (FHR) documented per mother
  • Number of times fetal heart rate (FHR) documented in labour
Intrapartum fetal monitoring - Improved documentation of fetal heart rate | 8 months
  Average time between last FHR documented and delivery (minutes)
  • Average time between last fetal heart rate (FHR) documented and delivery
Intrapartum fetal monitoring - Improved documentation (Risk factors for poor perinatal outcome) | 8 months
  Average number of fetal risk factors documented per mother
  • Risk factors for poor perinatal outcome
Intrapartum fetal monitoring - Cardiotocography (CTG) meetings | 8 months
  Average number of cases discussed per meeting
  • Number of cases (CTGs and poor perinatal outcomes) discussed
Training - number of staff trained | 8 months
  Number of staff trained as a percentage of the number of eligible staff. Senior doctors Residents Nurses/midwives Students
Training - Improvement in pre and post test scores | 8 months
  Percentage change between pre and post test scores, per staff member trained
Training - Improvement in self perceived knowledge and confidence about intrapartum fetal monitoring | 8 months
  Mean Likert score
Training - satisfaction and feedback about training | 8 months
  Survey data from staff attending training. Semi-structured questions.
Maternal - Caesarean section rate overall | 8 months
  Number of cases of caesarean section/month as a % of all births
Maternal - Operative vaginal delivery rate | 8 months
  Number of cases of operative delivery/month as a % of all births
Maternal - Maternal length of hospital stay | 8 months
  Average length of maternal stay/per patient/month
Maternal - Maternal death | 8 months
  Total number of maternal deaths/month
Perinatal - Apgar score | 8 months
  Number of cases of Apgar score 7 or below at 5 minutes/month as a percentage of all births
Perinatal - Cord blood lactate | 8 months
  Number of cases of cord blood lactate 4.9 mmol/l or above/month as a percentage of all births
Perinatal - Neonatal resuscitation | 8 months
  Number of babies requiring resuscitation/month as a percentage of all births
Perinatal - Neonatal intensive care unit (NICU) admission | 8 months
  Number of NICU admissions/month as a percentage of all births
Perinatal - Length of NICU stay | 8 months
  Average number of days/admission/month
Perinatal - Neonatal morbidity | 8 months
  Number of cases of birth asphyxia/HIE per month as a percentage of all births
Perinatal - Perinatal death before discharge | 8 months
  Number of perinatal deaths/month as a percentage of all births

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Weeks, Professor, Principal Investigator — University of Liverpool; Kate Lightly, Dr, Study Director — University of Liverpool
Locations (1):
- Government Medical College, Nagpur, Maharastra, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided